CLINICAL TRIAL: NCT07213804
Title: FRAmework-01: A Two-Part Phase 3 Study of Sofetabart Mipitecan (LY4170156) Versus Chemotherapy or Mirvetuximab Soravtansine in Platinum-Resistant Ovarian Cancer, and Sofetabart Mipitecan Plus Bevacizumab Versus Platinum-Based Chemotherapy Plus Bevacizumab in Platinum-Sensitive Ovarian Cancer.
Brief Title: A Two-Part Phase 3 Study of Sofetabart Mipitecan (LY4170156) in Participants With Platinum-Resistant (Part A) and Platinum-Sensitive (Part B) Ovarian Cancer
Acronym: FRAmework-01
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: GOG Foundation (Network); European Network of Gynaecological Oncological Trial Groups (ENGOT) (Other); Asia-Pacific Gynecologic Oncology Trials Group (APGOT) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 27727; 2025-522255-25-00 (EU CTIS Number); J5E-MC-JZXB (Other: Eli Lilly and Company); GOG-3133 (Other: Gynecologic Oncology Group); ENGOT-ov97/GINECO-NOGGO (Other: European Network of Gyneaecological Oncological Trial Groups); APGOT-OV17 (Other: Asia-Pacific Gynecologic Oncology Trials Group)
Record Dates: First submitted 2025-10-07; First posted 2025-10-09 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Ovarian Neoplasms; Fallopian Tube Neoplasms; Peritoneal Neoplasms; Neoplasm Metastasis
Keywords: Folate Receptor Alpha; Antibody-drug Conjugate; Platinum-Resistant; Platinum-Sensitive
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms; Peritoneal Neoplasms; Neoplasm Metastasis | interventions — Paclitaxel; Topotecan; Gemcitabine; liposomal doxorubicin; Bevacizumab; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part A: Sofetabart Mipitecan (Experimental): Administered intravenously (IV).
  Interventions: Drug: Sofetabart Mipitecan
- Part A: Chemotherapy or Mirvetuximab Soravtansine (MIRV) (Active Comparator): Investigator's Choice of Chemotherapy or MIRV given IV.
  Interventions: Drug: Paclitaxel; Drug: Topotecan; Drug: Gemcitabine; Drug: Pegylated liposomal doxorubicin (PLD); Drug: MIRV
- Part B: LY4170156 plus Bevacizumab (Experimental): Administered IV.
  Interventions: Drug: Sofetabart Mipitecan; Drug: Bevacizumab
- Part B: Platinum-based Doublet Chemotherapy plus Bevacizumab (Active Comparator): Investigator's choice of platinum doublet chemotherapy IV followed by bevacizumab IV.
  Interventions: Drug: Paclitaxel; Drug: Gemcitabine; Drug: Pegylated liposomal doxorubicin (PLD); Drug: Bevacizumab; Drug: Carboplatin

INTERVENTIONS:
Drug: Sofetabart Mipitecan — Administered IV
  Other Names: LY4170156
  Arms: Part A: Sofetabart Mipitecan; Part B: LY4170156 plus Bevacizumab
Drug: Paclitaxel — Administered IV
  Arms: Part A: Chemotherapy or Mirvetuximab Soravtansine (MIRV); Part B: Platinum-based Doublet Chemotherapy plus Bevacizumab
Drug: Topotecan — Administered IV
  Arms: Part A: Chemotherapy or Mirvetuximab Soravtansine (MIRV)
Drug: Gemcitabine — Administered IV
  Arms: Part A: Chemotherapy or Mirvetuximab Soravtansine (MIRV); Part B: Platinum-based Doublet Chemotherapy plus Bevacizumab
Drug: Pegylated liposomal doxorubicin (PLD) — Administered IV
  Arms: Part A: Chemotherapy or Mirvetuximab Soravtansine (MIRV); Part B: Platinum-based Doublet Chemotherapy plus Bevacizumab
Drug: MIRV — Administered IV
  Arms: Part A: Chemotherapy or Mirvetuximab Soravtansine (MIRV)
Drug: Bevacizumab — Administered IV
  Arms: Part B: LY4170156 plus Bevacizumab; Part B: Platinum-based Doublet Chemotherapy plus Bevacizumab
Drug: Carboplatin — Administered IV
  Arms: Part B: Platinum-based Doublet Chemotherapy plus Bevacizumab

SUMMARY:
This is a clinical study that has two parts. It is testing a potential new medicine called Sofetabart Mipitecan (LY4170156) for people with certain types of ovarian, peritoneal, and fallopian tube cancers. Part A looks at participants whose cancer no longer responds to platinum-based treatments (a type of chemotherapy). Part B looks at participants whose cancer still responds to platinum-based treatments. The researchers want to find out if Sofetabart Mipitecan works better than the usual treatments that doctors use now and to better understand how safe it is. Each participant's time in the study will depend on how they respond to the treatment.

ELIGIBILITY:
Inclusion Criteria:

Part A and B:

* Have histologically confirmed high-grade serous or high-grade endometrioid ovarian, primary peritoneal, or fallopian tube cancer.
* Have confirmed availability of tumor tissue block or slides
* Have radiographic progression on or after most recent line of systemic anticancer therapy
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
* Have measurable disease per RECIST v1.1

Part A:

* Have platinum-resistant disease, defined as radiographic progression less than or equal to (≤)6 months of the last administration of platinum therapy.
* Have previously received greater than or equal to (≥)1 but ≤3 prior lines of systemic cytotoxic therapy. Up to 4 lines of prior therapy is allowed if one of those lines is mirvetuximab soravtansine.
* Have received prior bevacizumab treatment, unless documented contraindication or intolerance.
* Have received treatment with a poly(ADP-ribose) polymerase inhibitor (PARPi) if known to have a somatic or germline breast cancer gene (BRCA) mutation, if clinically indicated, unless documented contraindication or intolerance.

Part B:

* Have relapsed after first-line platinum-based chemotherapy and have platinum-sensitive disease defined as radiographic progression greater than (>)6 months of their last administration of platinum therapy
* Have previously received ≥1 but ≤2 prior lines of systemic cytotoxic chemotherapy
* Have previously received a PARPi, per local product label, with progression on, or within 6 months of completion of PARPi treatment.

Exclusion Criteria:

Part A and B:

- Have received prior antibody-drug conjugate (ADC) with a topoisomerase inhibitor payload.

Part A:

- Have primary platinum-refractory disease, defined as disease that progressed ≤3 months since the last dose of first-line platinum-containing chemotherapy.

Part B:

- Have clinically significant proteinuria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1080 (Estimated)
Dates: Start 2025-10-22 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2031-08 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) | Randomization to radiographic progression or death from any cause (up to 70 months)
  PFS per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 by Investigator

SECONDARY OUTCOMES:
Overall Survival (OS) | Randomization to date of death from any cause (up to 70 months)
PFS | Randomization to radiographic progression or death from any cause (up to 70 months)
  PFS by blinded independent central review (BICR)
Overall Response Rate (ORR): Proportion of Participants who Achieve a Best Overall Response (BOR) of Complete Response (CR) or Partial Response (PR) | Randomization to disease progression or death (up to 70 months)
  ORR per RECIST v1.1
Duration of Response (DOR) | Date of first documented CR or PR to date of radiographic progression or death from any cause (up to 70 months)
  DOR per RECIST v1.1
Disease Control Rate (DCR): Proportion of Participants who Achieve a BOR of CR, PR, or Stable Disease (SD) | Randomization to disease progression or death from any cause (up to 70 months)
  DCR per RECIST v1.1
PFS2 | Randomization to disease progression on next line of treatment or death from any cause (up to 70 months)
Time to Initiation of First Subsequent Systemic Anticancer Therapy or Death (TNTD) | Randomization to initiation of subsequent systemic anticancer or death from any cause (up to 70 months)
Proportion of Participants with Response of Cancer Antigen-125 (CA-125) per Gynecologic Cancer Intergroup Criteria (GCIG) | Randomization to 30 days post treatment discontinuation
  Per GCIG
Percentage of Assessments with High Side-effect Bother, as measured by Functional Assessment of Cancer Therapy - General Item 5 (FACT GP5) | Randomization to 30 days post treatment discontinuation
  FACT-GP5 is a single-item, patient-reported instrument for assessing overall treatment side-effect burden. High side effect bother is defined as a score of 3 or 4 on a 5-point Likert scale. Higher scores represent higher symptom burden.
Change from Baseline in Abdominal/GI Symptoms, as measured by the European Organization for Research and Treatment of Cancer Ovarian Cancer Module (EORTC OV28) | Randomization to 30 days post treatment discontinuation
  The EORTC OV28 consists of 28 items covering 3 functional scales and 5 symptom scales. The Abdominal/GI symptom scale ranges from 0 to 100. Higher scores indicate worse symptoms.
Change from Baseline in Overall Health-related Quality of Life (HRQoL), as measured by the EORTC QLQ-C30 Global Health Status/Quality of Life Subscale | Randomization to 30 days post treatment discontinuation
  The EORTC QLQ-C30 is a 30-question patient-reported instrument used to assess multidimensional HRQoL in cancer patients. Overall HRQoL is measured by the EORTC QLQ-30 Global Health Status/Quality of Life Subscale (two items). Response options range from 0 - 100. Higher score represents better overall HRQoL.
Pharmacokinetics (PK): Minimum Blood Plasma Concentration (Cmin) of LY4170156 | Randomization through end of treatment (up to 70 months)]

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (245):
- United States (76):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - HonorHealth, Phoenix, Arizona
  - Roy and Patricia Disney Family Cancer Center - Providence Saint Joseph Medical Center, Burbank, California
  - Moores Cancer Center, La Jolla, California
  - UCLA Hematology/Oncology - Westwood (Building 100), Los Angeles, California
  - Stanford Women's Cancer Center, Palo Alto, California
  - Kaiser Permanente Zion Medical Center, San Diego, California
  - Sansum Clinic, Solvang, California
  - Kaiser Permanente, Vallejo, California
  - Anschutz Cancer Pavilion, Aurora, Colorado
  - AdventHealth Medical Group - Porter, Denver, Colorado
  - UConn Health, Farmington, Connecticut
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Florida Cancer Specialist- South, Fort Myers, Florida
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - University of Miami Hospital and Clinics, Sylvester Cancer Center, Miami, Florida
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Florida Cancer Specialist- East, West Palm Beach, Florida
  - Nancy N. & J.C. Lewis Cancer and Research Pavillion, Savannah, Georgia
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Illinois Cancer Specialists, Arlington Heights, Illinois
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - OSF Saint Fracis Medical Center, Peoria, Illinois
  - Franciscan Health, Indianapolis, Indiana
  - Baptist Health Lexington, Lexington, Kentucky
  - Norton Women's and Children's Hospital, Louisville, Kentucky
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Trials 365, Shreveport, Louisiana
  - Maine Medical Center - Scarborough Campus, Scarborough, Maine
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Sinai Hospital Of Baltimore, Baltimore, Maryland
  - University of Massachusetts Chan Medical School, Worcester, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Mayo Clinic in Rochester, Minnesota, Rochester, Minnesota
  - University of Missouri Hospital, Columbia, Missouri
  - Cox Medical Center North, Springfield, Missouri
  - The Center of Hope, Reno, Nevada
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Holy Name Medical Center, Teaneck, New Jersey
  - Optimum Clinical Research Group, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Northwell Health/ RJ Zuckerberg Cancer Center, Lake Success, New York
  - Perlmutter Cancer Center at NYU Langone Hospital - Long Island, Mineola, New York
  - Laura and Isaac Perlmutter Cancer Center, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - Duke Cancer Institute, Durham, North Carolina
  - Miami Valley Hospital South, Centerville, Ohio
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Oncology Hematology Care Inc, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - The James Cancer Hospital and Solove Research Institute at The Ohio State University Comprehensive Cancer -T, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - USO - Oncology Associates of Oregon, P. C., Eugene, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Kaiser Permanente Interstate Medical Office Central, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - University of Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Asplundh Cancer Pavilion, Willow Grove, Pennsylvania
  - Women & Infants Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - USO-Texas Oncology-Central/South Texas, Austin, Texas
  - US Oncology, The Woodlands, Texas
  - USO - Texas Oncology Gulf Coast, Webster, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Swedish Cancer Institute - Edmonds, Edmonds, Washington
  - Swedish Medical Center, Seattle, Washington
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
- Australia (5):
  - Ballarat Health Services, Ballarat Central
  - Gold Coast University Hospital, Southport
  - Royal North Shore Hospital, St Leonards
  - The Townsville Hospital, Townsville
  - Latrobe Regional Health, Traralgon
- Austria (3):
  - Medizinische Universität Graz, Graz
  - Medizinische Universitaet Innsbruck, Innsbruck
  - Universitaetsklinikum Allgemeines Krankenhaus Wien, Vienna
- Belgium (5):
  - Institut Jules Bordet, Anderlecht
  - AZ Sint-Jan Brugge-Oostende AV, Bruges
  - Antwerp University Hospital, Edegem
  - AZ Maria Middelares, Ghent
  - UZ Leuven, Leuven
- Brazil (8):
  - CPAM - Centro de Pesquisas da Amazônia, Belém
  - Oncocentro de Minas Gerais, Belo Horizonte
  - CEPEN - Centro de Pesquisa e Ensino em Oncologia de Santa Catarina, Florianópolis
  - Hospital Brasilia, Lago Sul
  - Centro de Tratamento de Tumores Botafogo para Oncoclinicas Rio de Janeiro SA, Rio de Janeiro
  - Instituto D'Or Pesquisa e Ensino, Rio de Janeiro
  - Clinica Amo - Rio Vermelho, Salvador
  - Centro de Oncologia - CEON+ - Unidade São Caetano do Sul, São Caetano do Sul
- Canada (7):
  - Arthur J.E. Child Comprehensive Cancer Centre, Calgary
  - Hamilton Health Sciences-Juravinski Cancer Centre, Hamilton
  - Jewish General Hospital, Montreal
  - Centre intégré universitaire de santé et de services sociaux de l'Estrie Centre Hospitalier Universitaire -T, Sherbrooke
  - BC Cancer Surrey, Surrey
  - Sunnybrook Research Institute, Toronto
  - Princess Margaret Cancer Centre, Toronto
- China (25):
  - Peking University First Hospital, Beijing
  - Beijing Cancer hospital, Beijing
  - The First Hospital of Jilin University, Changchun
  - The First People's Hospital of Changde City, Changde
  - Xiangya Hospital Central South University, Changsha
  - West China Second University Hospital, Sichuan University, Chengdu
  - Fujian Cancer Hospital, Fuzhou
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou
  - Zhujiang Hospital, Guangzhou
  - Sun Yat-Sen University Cancer Centre, Guangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Shandong Cancer Hospital, Jinan
  - Gansu Provincial Maternity and Child Care Hospital, Lanzhou
  - The First Affiliated Hospital of Henan University of Science &Technology, Luoyang
  - Nanjing Drum Tower Hospital The Affiliated Hospital of Nanjing University Medical School, Nanjing
  - Jiangsu Province Hospital, Nanjing
  - Guangxi Medical University Affiliated Tumor Hospital, Nanning
  - Obstetrics & Gynecology Hospital of Fudan University, Shanghai
  - Fudan University Shanghai Cancer Center, Shanghai
  - Cancer Hospital of Shantou University Medical College, Shantou
  - Peking University Shenzhen Hospital, Shenzhen
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin
  - Wuhan Union Hospital, Wuhan
  - Tongji Hospital, Tongji Medical College of Huazhong University of Science and Technology, Wuhan
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an
- Czechia (5):
  - Fakultní Nemocnice Brno, Brno
  - Nemocnice AGEL Novy Jicin a.s., Nový Jiín
  - Fakultni nemocnice Olomouc, Olomouc
  - Vseobecna fakultni nemocnice v Praze, Prague
  - Nemocnice Tomase Bati ve Zline, Zlín
- Denmark (2):
  - Rigshospitalet, Copenhagen
  - Vejle Sygehus, Vejle
- France (11):
  - Institut de Cancérologie de l'Ouest, Angers
  - Centre Hospitalier de la Côte Basque, Bayonne
  - Institut Bergonié - Centre Régional de Lutte Contre Le Cancer de Bordeaux et Sud Ouest, Bordeaux
  - CHRU de Brest, Brest
  - Centre Oscar Lambret, Lille
  - Centre Hospitalier Universitaire de Limoges - Hôpital Dupuytren, Limoges
  - Centre Leon Berard, Lyon Cedex08
  - Institut Régional du Cancer Montpellier, Montpellier
  - Hopitaux Universitaires Paris Centre-Hopital Cochin, Paris
  - Groupe Hospitalier Diaconesses Croix Saint Simon, Paris
  - CHU Strasbourg-Hautepierre, Strasbourg
- Germany (9):
  - Universitätsklinikum Aachen, Aachen
  - Charité Campus Virchow-Klinikum, Berlin
  - Universitätsklinikum Bonn, Bonn
  - Universitaetsklinikum Koeln, Cologne
  - Universitaetsklinikum Carl Gustav Carus Dresden, Dresden
  - Universitaetsklinikum Duesseldorf, Düsseldorf
  - Universitaetsklinikum Erlangen, Erlangen
  - Kliniken Essen-Mitte, Evangelische Huyssens-Stiftung, Essen
  - Universitaetsklinikum Schleswig-Holstein Campus Kiel, Kiel
- Greece (4):
  - Alexandra Hospital, Athens
  - Aretaieio Hospital, Athens
  - General Hospital of Kalamata, Kalamata
  - General Oncology Hospital of Kifissia "Agioi Anargiroi", Nea Kifissia
- Hungary (2):
  - Országos Onkológiai Intézet, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
- Ireland (3):
  - Cork University Hospital, Cork
  - St. Vincent's University Hospital, Dublin
  - St. James's Hospital, Dublin
- Italy (12):
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna, Policlinico di Sant'Orsola, Bologna
  - Ospedale Cannizzaro, Catania
  - Ospedale Vito Fazzi, Lecce
  - Azienda USL 2 Lucca, Lucca
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Istituto Europeo di Oncologia IRCCS, Milan
  - Ospedale Humanitas San Pio X, Milan
  - Azienda Ospedaliero Universitaria, Modena
  - Istituto Nazionale Tumori IRCCS Fondazione Pascale, Napoli
  - Nuovo Ospedale di Prato-S.Stefano, Prato
  - Ospedale Santa Maria delle Croci, Ravenna
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS - Università Cattolica del Sacro Cuore, Roma
- Japan (15):
  - Hyogo Cancer Center, Akashi
  - National Cancer Center Hospital, Chūōku
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - Saitama Medical University International Medical Center, Hidaka
  - National Cancer Center Hospital East, Kashiwa
  - The Cancer Institute Hospital of JFCR, Kōtoku
  - Nagoya University Hospital, Nagoya
  - Niigata Cancer Center Hospital, Niigata
  - Okayama University Hospital, Okayama
  - Hokkaido University Hospital, Sapporo
  - Tohoku University Hospital, Sendai
  - Iwate Medical University Hospital, Shiwa-gun Yahaba-cho
  - The University of Osaka Hospital, Suita
  - Ehime University Hospital, Tōon
  - Mie University Hospital, Tsu
- Mexico (6):
  - Scientia Investigacion Clinica S.C., Chihuahua City
  - Health Pharma Professional Research S.A. de C.V:, Mexico City
  - Higiea Oncologia, Mexico City
  - INCAN, Mexico City
  - Unidad Médica Onco-hematológica, Puebla City
  - Hospital Angeles, Tijuana
- Netherlands (2):
  - University Medical Center Groningen, Groningen
  - Erasmus Medisch Centrum, Rotterdam
- Norway (2):
  - Oslo universitetssykehus, Radiumhospitalet, Oslo
  - Stavanger Universitetssykehus, Stavanger
- Poland (5):
  - Uniwersytecki Szpital Kliniczny w Białymstoku, Bialystok
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - SP ZOZ Szpital Uniwersytecki w Krakowie, Krakow
  - Wielkopolskie Centrum Onkologii im. Marii Skłodowskiej-Curie, Poznan
  - Mazowiecki Szpital Wojewódzki w Siedlcach, Siedlce
- Romania (4):
  - SC Memorial Healthcare International SRL, Bucharest
  - Sc Mnt Healthcare Europe Srl, Bucharest
  - Institutul Regional de Oncologie, Iași
  - S C Oncocenter Oncologie Clinica S R L, Timișoara
- South Korea (8):
  - Keimyung University Dongsan Hospital, Daegu
  - National Cancer Center, Goyang-si
  - Seoul National University Bundang Hospital, Seongnam
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Ajou University Hospital, Suwon
- Spain (8):
  - Hospital Universitari Dexeus, Barcelona
  - Hospital Provincial Centre de Castelló, Castellon
  - Hospital Universitario Virgen Nieves, Granada
  - Hospital Universitario HM Sanchinarro, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario Infanta Sofía, San Sebastián de los Reyes
  - CHUS - Hospital Clinico Universitario, Santiago de Compostela
  - Hospital Universitario de Toledo, Toledo
- Switzerland (4):
  - Kantonsspital Baden, Baden
  - Ospedale Regionale Bellinzona e Valli, Bellinzona
  - Kantonsspital Graubünden, Chur
  - Hôpitaux Universitaires de Genève (HUG), Geneva
- Taiwan (8):
  - Chang Gung Memorial Hospital at Kaohsiung, Kaohsiung Niao Sung Dist
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Mackay Memorial Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Medical Foundation-Linkou Branch, Taoyuan District
- United Kingdom (6):
  - Royal United Hospitals NHS Foundation Trust, Bath
  - St James's University Hospital, Leeds
  - Royal Marsden Hospital (Sutton), London
  - Royal Marsden Hospital (Chelsea), London
  - The Christie NHS Foundation Trust, Manchester
  - Torbay Hospital, Torquay

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication or approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal should be approved by an independent review panel and researchers should sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- See also: Related Info — https://trials.lilly.com/en-US/trial/660615